CLINICAL TRIAL: NCT01034943
Title: Dorsally Displaced Extraarticular Distal Radius Fractures - Volar Plate or External Fixation. A Prospective Randomized Trial
Brief Title: Extraarticular Distal Radius Fractures, X-fix or Volar Fixation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Sari Ponzer, Professor, MD, Consultant orthopeadic surgeon, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRF Extra
Record Dates: First submitted 2009-12-16; First posted 2009-12-18 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Dorsally Displaced Intraarticular Distal Radius Fractures; Age 50 - 74 for Females or 60-74 for Males; Low Energy Trauma
Keywords: radius; fracture; wrist; external; fixation; volar; plate; DASH; PRWE
MeSH Terms: conditions — Fractures, Bone | interventions — External Fixators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- External fixation (Active Comparator): Operation with external fixation and optional addition of k-wire
  Interventions: Procedure: External fixation
- Volar plate (Active Comparator): Operation with Synthes volar two column plate (TCP)
  Interventions: Procedure: Volar plate

INTERVENTIONS:
Procedure: External fixation — Operation with external fixation and optional addition of k-wire
  Other Names: External Fixation with Hoffman external fixator (Stryker)
  Arms: External fixation
Procedure: Volar plate — Operation with a Synthes volar two column plate (TCP)
  Other Names: Synthes volar two column plate (TCP)
  Arms: Volar plate

SUMMARY:
Distal radius fractures are treated surgically if severely displaced. This study aims to investigate the outcome after surgery. The investigators will randomize patients to either external fixation with optional addition of k-wires or open reduction and fixation with a volar plate.

DETAILED DESCRIPTION:
This study has been merged with study NCT01035359 and a new ethical permission has been granted by the Swedish National Ethic board

ELIGIBILITY:
Inclusion Criteria:

* Female 50-74 years or male 60-74 years
* Dorsally displaced extraarticular distal radius fracture
* Dorsal angulation >20 degrees measured from the plane perpendicular to the radius axis
* Low energy trauma
* Injury <72 hours when diagnosed
* Patient independent of help for ADL

Exclusion Criteria:

* Earlier dysfunction in any wrist
* Other major injuries
* Rheumatoid arthritis or other systemic joint disease
* Dementia or severe psychiatric disease
* Severe medical condition making general anesthesia a considerable risk

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-08; Primary Completion 2013-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome is measured by DASH (Disability of the Arm, Shoulder and Hand), which is a self administered questionnaire validated for disease and dysfunction of the upper limb. | 12 months

SECONDARY OUTCOMES:
A secondary outcome measure is the degree of malalignment on the x-ray of the injured wrist. | 12 months
A secondary outcome measure for this study is the EQ5D, a validated quality-of-life instrument. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sari Ponzer, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Stockholm South Hospital Department of Orthopeadic Surgery, Stockholm, Stockholm County, Sweden